CLINICAL TRIAL: NCT01215734
Title: Randomized Double-Blind, Comparison of Standard Dose Trivalent Inactivated Influenza Vaccine Versus High-Dose Trivalent Inactivated Influenza Vaccine in Adult Stem Cell Hematopoetic Transplant Recipients
Brief Title: Standard vs High-Dose Trivalent Inactivated Flu Vaccine in Adult Hematopoetic Stem Cell Transplant (HSCT) Recipients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Natasha Halasa, MD, Assistant Professor of Pediatrics, Pediatric Infectious Diseases, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VICC BMT 1057; 100980 (Other: IRB number); 100980 (Other: IRB number, no grant for this study)
Record Dates: First submitted 2010-10-05; First posted 2010-10-06 (Estimated); Results first posted 2013-03-08 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-02

CONDITIONS: Adult Stem Cell Hematopoetic Transplant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High-Dose Trivalent Inactivated Influenza Vaccine (Active Comparator): Forty adult hematopoetic stem cell transplant recipients at least 6 months post transplant will receive high dose trivalent influenza vaccine
  Interventions: Biological: High-Dose Trivalent Inactivated Influenza Vaccine (HD-TIV)
- Standard dose Trivalent Inactivated Flu Vaccine (Active Comparator): Twenty Adult stem cell transplant recipients at least 6 months post transplant will receive standard dose trivalent influenza vaccine.
  Interventions: Biological: Standard Dose Trivalent Inactivated Flu Vaccine

INTERVENTIONS:
Biological: High-Dose Trivalent Inactivated Influenza Vaccine (HD-TIV) — 0.5 ml of HD-TIV on visit 1
  Arms: High-Dose Trivalent Inactivated Influenza Vaccine
Biological: Standard Dose Trivalent Inactivated Flu Vaccine — Twenty adult hematopoetic stem cell transplant recipients will receive 0.5 ml standard dose trivalent influenza vaccine on visit 1.
  Arms: Standard dose Trivalent Inactivated Flu Vaccine

SUMMARY:
Hypothesis 1: The safety profile in adult allogeneic stem cell hematopoietic transplant (SCT) recipients after high dose (HD) trivalent inactivated influenza vaccine (TIV) will not be significantly different from adult stem cell transplant recipients receiving standard dose (SD) TIV.

* Specific Aim 1: To compare safety profile of high dose trivalent inactivated influenza vaccine to standard dose trivalent inactivated influenza vaccine in adult hematopoietic stem cell transplant recipients.

Hypothesis 2: Adult stem cell transplant recipients who received the higher dose trivalent influenza vaccine will have a greater frequency of (at least a 4-fold) rise in antibody titers to influenza antigens compared to those who receive standard dose trivalent influenza vaccine.

* Specific Aim 2: To compare humoral immune responses of adult hematopoietic stem cell transplant recipients influenza virus antigens included in trivalent influenza vaccine after high dose or standard dose trivalent influenza vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Allogeneic hematopoietic stem cell transplant recipients who are >6 post-transplant
* greater than or equal to 18 years of age
* Available for duration of study
* If patients are on immunosuppressive therapy for treatment of graft versus host disease (GVHD): only those on stable doses for at least 4 weeks or on tapering doses will be eligible.

Exclusion Criteria:

* History of hypersensitivity to previous influenza vaccination or hypersensitivity to eggs/egg protein
* History of Guillain-Barre syndrome
* Evidence of hematologic malignancy or disease relapse post-transplant (mixed chimerisms and molecular evidence of disease is permitted)
* Non-allogeneic (e.g. autologous) hematopoietic SCT recipients
* History of receiving 2011 - 2012 influenza vaccine
* History of proven influenza disease after September 1, 2011.
* Pregnant females
* Have any condition that would, in the opinion of the site investigator, place them at an unacceptable risk of injury or render them unable to meet the requirements of the protocol
* Have any condition that the investigator believes may interfere with successful completion of the study
* Platelet count less than 50,000 cells/μL
* History of known infection with HIV, Hepatitis B or Hepatitis C
* History of known latex hypersensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Halasa, M.D., M.P.H., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt-Ingram Cancer Center, Clinical Trials Information Program, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This phase X, double-blind study was conducted from September 2011 - April 2012.
Pre-assignment Details: Forty-seven patients consented to participate in this study, three were determined ineligible.
Groups:
- High-Dose Trivalent Inactivated Influenza Vaccine: Forty adult hematopoetic stem cell transplant recipients at least 6 months post-transplant will receive high dose trivalent influenza vaccine
  High-Dose Trivalent Inactivated Influenza Vaccine (HD-TIV) : 0.5 ml of HD-TIV on visit 1
- Standard Dose Trivalent Inactivated Flu Vaccine: Twenty Adult stem cell transplant recipients at least 6 months post-transplant will receive standard dose trivalent influenza vaccine.
  Standard Dose Trivalent Inactivated Flu Vaccine : Twenty adult hematopoetic stem cell transplant recipients will receive 0.5 ml standard dose trivalent influenza vaccine on visit 1.
Period: Overall Study
Arm/Group | High-Dose Trivalent Inactivated Influenza Vaccine | Standard Dose Trivalent Inactivated Flu Vaccine
Started | 29 | 15
Completed | 29 | 14
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-Dose Trivalent Inactivated Influenza Vaccine | Standard Dose Trivalent Inactivated Flu Vaccine | Total
Number analyzed (Participants) | 29 | 15 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 14 | 41
  >=65 years | 2 | 1 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 50 (12) | 49 (14) | 50 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 5 | 16
  Male | 18 | 10 | 28
Region of Enrollment [Number; unit: participants]
  United States | 29 | 15 | 44

OUTCOME MEASURES:

1. Primary Outcome: Patients Experiencing at Least 1 Solicited Local and/or Systemic Adverse Event After High Dose (HD) Trivalent Influenza Vaccine (TIV) or Standard Dose (SD) Trivalent Influenza Vaccine in Adult Hematopoetic Stem Cell Transplant (SCT) Recipients
Description: Patients were questioned about the following adverse events related to TIV: Local: pain, tenderness, swelling/induration, or erythema at injection site. Systemic: fatigue/malaise, headache, nausea, vomiting, body ache not at injection site, fever >= 100.4 degrees Fahrenheit, or change in activity level.
Time Frame: Day of TIV to 7 days after TIV
Population: Patients who received either the high-dose TIV or the standard dose TIV
Measure: Number; unit: participants
Groups:
- High-Dose Trivalent Inactivated Influenza Vaccine: High Dose: Adult hematopoetic stem cell transplant recipients at least 6 months post transplant will receive HD TIV (60 micrograms [µg] per antigen) on visit 1
- Standard Dose Trivalent Inactivated Flu Vaccine: Standard Dose TIV : Adult hematopoetic stem cell transplant recipients at least 6 months post-transplant will receive SD (15 µg/per antigen) TIV on visit 1.
Arm/Group | High-Dose Trivalent Inactivated Influenza Vaccine | Standard Dose Trivalent Inactivated Flu Vaccine
Number analyzed (Participants) | 29 | 15
participants
  Local Adverse Events | 18 | 4
  Systemic Adverse Events | 14 | 7

2. Secondary Outcome: Patients Receiving HD or SD TIV With a 4-fold Rise in Hemagglutination Inhibition (HAI) Titers Relative to Baseline for Each of 3 Influenza Viruses
Description: Adult hematopoetic stem cell transplant recipients at least 6 months post-transplant receiving either HD or SD TIV who had blood drawn at pre-vaccination and at 28-42 days post-vaccination and who experienced a 4-fold rise in each of three post-vaccination influenza antibody titers, relative to their baseline titers. Trivalent vaccine is for the H1N1/H3N2/B influenzas. A 4-fold rise in type-specific antibody titer is considered adequate antibody response to the specific influenza virus
Time Frame: Before TIV and 28-42 days after TIV
Population: Patients who received either the high-dose or the standard dose TIV and who had blood drawn for HAI titers before TIV and at 28-42 days after TIV. Data not available for 5 HD and 1 SD patients.
Measure: Number; unit: participants
Arm/Group | High-Dose Trivalent Inactivated Influenza Vaccine | Standard Dose Trivalent Inactivated Flu Vaccine
Number analyzed (Participants) | 24 | 14
participants
  H1N1 Influenza | 12 | 5
  H3N2 Influenza | 10 | 5
  B Influenza | 10 | 6

ADVERSE EVENTS:
Groups:
- High-Dose Trivalent Inactivated Influenza Vaccine: Forty adult hematopoetic stem cell transplant recipients at least 6 months post transplant will receive high dose trivalent influenza vaccine
  High-Dose Trivalent Inactivated Influenza Vaccine (HD-TIV) : 0.5 ml of HD-TIV on visit 1
- Standard Dose Trivalent Inactivated Flu Vaccine: Twenty Adult stem cell transplant recipients at least 6 months post transplant will receive standard dose trivalent influenza vaccine.
  Standard Dose Trivalent Inactivated Flu Vaccine : Twenty adult hematopoetic stem cell transplant recipients will receive 0.5 ml standard dose trivalent influenza vaccine on visit 1.
Arm/Group | High-Dose Trivalent Inactivated Influenza Vaccine | Standard Dose Trivalent Inactivated Flu Vaccine
Serious Adverse Events (participants affected / at risk) | 11/29 | 7/15
Other Adverse Events (participants affected / at risk) | 5/29 | 5/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Dose Trivalent Inactivated Influenza Vaccine (N=29) | Standard Dose Trivalent Inactivated Flu Vaccine (N=15)
fever (General disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
chest pain, cardiac (Cardiac disorders) | 0 (0) | 1 (2)
heart failure (Cardiac disorders) | 1 (1) | 0 (0)
palpitations (Cardiac disorders) | 0 (0) | 1 (1)
pericardial effusion (Cardiac disorders) | 1 (2) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
malaise (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Infections and infestations other (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
weight loss (Investigations) | 1 (1) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Planned knee replacement surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chronic inflammatory demyelinating polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
bonchitis obliterans (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Methicillin-resistant Staphylococcus aureus bacteremia (Infections and infestations) | 0 (0) | 1 (1)
rectal abscess (Gastrointestinal disorders) | 1 (1) | 0 (0)
diffuse muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-Dose Trivalent Inactivated Influenza Vaccine (N=29) | Standard Dose Trivalent Inactivated Flu Vaccine (N=15)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
investigations, other (Investigations) | 2 (2) | 1 (1)
anorexia (Gastrointestinal disorders) | 2 (2) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
edema limbs (General disorders) | 0 (0) | 1 (1)
hepatobiliary disorders, other (Hepatobiliary disorders) | 0 (0) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
mucositits oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
skin and other subcutaneous disorders-other (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes